CLINICAL TRIAL: NCT05857696
Title: Study of the Improvement of Gait by Spinal Stimulation in Patients With Post-operative Chronic Lumbosciatalgia: Pilot Study
Brief Title: Improvement of Gait by Spinal Stimulation in Patients With Postoperative Chronic Lumbosciatalgia: Pilot Study (GaitStim)
Acronym: GAITSTIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-AOI-09
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Failed Back Surgery Syndrome
Keywords: Spinal cord neurostimulation; chronic pain
MeSH Terms: conditions — Failed Back Surgery Syndrome; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Prospective study on the evolution of spatial-temporal parameters of walking for each mode of medullary neurostimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neurostimulation (Other): 3 months of tonic stimutaltion + 3 weeks with random stimulation mode between microburst, High frequency, stopped stimulation (Off) then stimulation with the more efficient mode (according the patient) until 6 monthe after implantation.
  Interventions: Other: walking quantified analysis

INTERVENTIONS:
Other: walking quantified analysis — Test to measure anthropometry, joint amplitudes, muscle strength and spasticity of the lower limbs on a treadmill.

SUMMARY:
The purpose of this study is to explore the changes in objective walking parameters induced by medullary stimulation in patients with Fail Back Surgery Syndrome, after chronic stimulation, in comparison with preoperative condition.

DETAILED DESCRIPTION:
After the informed consent signature, a first assessment will be carried out, including: quantified analysis of walking (AQM), felt effort questionnaire, pain questionnaires, functional abilities, limitations, goals and quality of life.

The implantation of the spinal cord stimulation system will be performed in two stages: the first stage, the electrode alone will be implanted and connected to an external test stimulator, allowing a one-week stimulation test.

If the test is positive (EVA pain improvement > or = 50%), the second step will be to connect this electrode to a Spectra WaveWriter™ internal stimulator. This stimulator delivers three different stimulation modalities: tonic, microburst and high frequency. The activated initial stimulation mode will be the tonic one.

After 3 months of "tonic" stimulation, the patient will be treated successively and in random way by 3 other different stimulation modalities during a week: microburst, high frequency, stopped stimulation (Off). The AQM and the different questionnaires will be done again, which will determine which stimulation modality is most beneficial to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year old and < or = 70 year old
* Patients with chronic neuropathic lumbo-sciatalgia (DN4 score > or = 4/10) as part of a moderate to severe spinal surgery failure syndrome (EVA >50/100), in who a collegial and multidisciplinary indication of medullary stimulation treatment was chosen.
* Patients awith Social Security

Exclusion Criteria:

* Vulnerable persons
* Patients who are invalid and unable to perform a quantified walk analysis
* Contraindication to surgery or anesthesia
* Patient not able to complete questionnaires
* Woman of childbearing age without effective contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
To explore the changes in objective walking parameters induced by spinal stimulation in patients with FBSS, after 6 months of chronic stimulation, in comparison with preoperative status. | At baseline, 3 and 6 months after implantation
  Gait quantified analysis with Gait Deviation Index

SECONDARY OUTCOMES:
To describe the gait alteration in a population of patients with FBSS | At baseline, 3 and 6 months after implantation
  Gait quantified analysis with Gait Deviation Index

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No